CLINICAL TRIAL: NCT03088085
Title: The Effectiveness of Self-thoracic Spine Mobilization on Improving Sleep Quality in Patients Who Have Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 092016-072
Record Dates: First submitted 2017-03-08; First posted 2017-03-23 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Shoulder Pain Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-mobilization (Experimental): Use of foam roller to mobilize thoracic spine and ribs every night before going to bed
  Interventions: Procedure: Self-mobilization
- Sleep Education (Active Comparator): Education on sleep hygiene with tips for improving sleep.
  Interventions: Procedure: Sleep Education

INTERVENTIONS:
Procedure: Self-mobilization — Subjects will mobilize thoracic spine and ribs with a foam roller every night before going to bed.
  Arms: Self-mobilization
Procedure: Sleep Education — Subjects will be educated on sleep hygiene in order to improve likelihood of having good sleep.
  Arms: Sleep Education

SUMMARY:
This project aims to study the impacts of self-thoracic spine and rib mobilization on sleep quality in patients who present to UTSW physicians with shoulder pain. The investigators plan to randomize participants into treatment and control groups, but the investigators will provide education on sleep hygiene for each group. The treatment group will also receive instruction to mobilize their thoracic spine and ribs each night before going to sleep.

DETAILED DESCRIPTION:
Subjects with a chief complaint of musculoskeletal pain will be recruited from clinics in the Departments of Internal Medicine, Family Medicine, and Orthopedic Surgery. Subjects will be randomized into either the intervention or control group. The intervention group will receive education on sleep hygiene and instruction to use a foam roller to mobilize the thoracic spine and ribs just before the subject goes to sleep. The control group will receive education on sleep hygiene. Valid and reliable measures will be used to assess sleep quality (Pittsburgh Sleep Quality Index), pain (Numeric Pain Rating Scale), and function (SF-36 and ASES), as well as a sleep diary. Measures will be taken at baseline as well as two weeks after the subject's enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain with associated sleeping disturbance
* Between the ages of 18-89
* Present to the clinics in the Departments of Internal Medicine, Family Medicine, and Orthopedic Surgery at UTSW

Exclusion Criteria:

* non-English speakers
* chronic pain or rheumatic disorders
* unstable psychopathology, cognitive impairment (including dementia)
* current or recent history (within 6 months) of substance abuse disorders
* recent history of surgery or fracture to the cervical spine, thoracic spine, ribs, or shoulders (within 6 months)
* metabolic bone disease (including osteoporosis)
* fusion or ankyloses
* osteomyelitis, pregnancy, vertebral basilar insufficiency, neoplastic disease, malignancy in the area of treatment
* actively treated for sleep disorders (including insomnia)
* uncontrolled congestive heart failure, COPD, hypertension, or other serious medical illness

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Index | Baseline, 1 week, and 2 weeks
  Valid and reliable 19 item assessment of sleep quality, with higher scores indicating greater sleep disturbance

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | Baseline, 1 week, and 2 weeks
  Valid and reliable 11 point rating of pain, with higher scores indicating more pain
SF-36 | Baseline, 1 week, and 2 weeks
  Valid and reliable 36 item assessment of quality of life, with higher scores indicating lower disability

CONTACTS AND LOCATIONS:
Overall Officials: Tara Dickson, DPT, Principal Investigator — Assistant Professor
Locations (1):
- Health Professions Physical Therapy Clinic, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No